CLINICAL TRIAL: NCT07062913
Title: Effectiveness of Contrast Compression Therapy for Post-Stroke Complex Regional Pain Syndrome: A Randomized Control Trial
Brief Title: Contrast Compression Therapy for Post-Stroke Complex Regional Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meltem Gunes Akinci (Other)
Responsible Party: Sponsor-Investigator, Meltem Gunes Akinci, Assistant Professor of Physical Medicine and Rehabilitation, Pamukkale University
Organization: Pamukkale University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E2-21-527
Record Dates: First submitted 2025-07-03; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Stroke; Complex Regional Pain Syndrome; Hemiplegia
Keywords: Stroke; Complex Regional Pain Syndrome; Contrast Compression Therapy; Hemiplegia; Neurorehabilitation
MeSH Terms: conditions — Stroke; Complex Regional Pain Syndromes; Hemiplegia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Rehabilitation Group (Active Comparator)
  Interventions: Procedure: Conventional Rehabilitation
- Contrast Compression Therapy Group (Experimental)
  Interventions: Device: Contrast Compression Therapy; Procedure: Conventional Rehabilitation

INTERVENTIONS:
Procedure: Conventional Rehabilitation — A standard rehabilitation program including positioning, range of motion exercises, stretching, strengthening, and conventional transcutaneous electrical nerve stimulation.
  Arms: Conventional Rehabilitation Group
Device: Contrast Compression Therapy — Contrast compression therapy using a Game Ready® MED4 ELITE device applied to the affected upper extremity with sequential hot and cold phases and pneumatic compression.
  Arms: Contrast Compression Therapy Group
Procedure: Conventional Rehabilitation — Same standard rehabilitation program as in the control group.
  Arms: Contrast Compression Therapy Group

SUMMARY:
This study aims to evaluate the effectiveness of contrast compression therapy as an adjunct to conventional rehabilitation in patients diagnosed with complex regional pain syndrome (CRPS) following stroke. Post-stroke CRPS, previously known as shoulder-hand syndrome, is a challenging condition that affects upper extremity function and quality of life. Although various conservative treatments such as medication, physical therapy, and contrast water therapy have been used with varying success, evidence for standardized protocols remains limited.

In this prospective, single-center, single-blind, randomized controlled trial, eligible patients with post-stroke CRPS type I were randomly assigned to receive either conventional rehabilitation alone or combined with contrast compression therapy. The intervention included 10 sessions of sequential thermal phases with pneumatic compression applied to the affected upper limb, delivered with a specialized device in addition to standard therapy.

The primary outcome measures were pain level and edema volume. Secondary outcomes included functional recovery, spasticity, clinical motor recovery, and neuropathic pain assessments. This study aims to contribute new evidence about whether contrast compression therapy offers additional benefits for managing post-stroke CRPS.*

DETAILED DESCRIPTION:
Post-stroke complex regional pain syndrome (CRPS), also known as shoulder-hand syndrome, is observed in more than 50% of patients who have experienced a stroke. This condition is typically classified as Type I CRPS due to the absence of identifiable peripheral nerve injury. Although the precise underlying mechanism remains unclear, biomechanical factors that cause mechanical instability of the shoulder joint and repetitive microtrauma are considered major risk factors for its development.

Clinically, post-stroke CRPS is characterized by severe pain involving both the shoulder and wrist, accompanied by symptoms such as edema, warmth, redness, limited range of motion, tenderness in the metacarpophalangeal joints, and in later stages, joint contractures that may cause significant functional impairment. The chronic nature of CRPS can lead to substantial limitations in upper extremity use, prolonged hospital stays, dependency in daily living activities, and increased overall rehabilitation costs, thereby reducing patients' quality of life.

Although various conservative treatments-including pharmacological agents, physical therapy, contrast water therapy (CWT), and sympathetic nerve blocks-are frequently used, the effectiveness, long-term safety, and accessibility of standardized treatment protocols remain limited. Traditional contrast water therapy aims to stimulate circulation and modulate inflammation by alternating vasodilation and vasoconstriction phases; however, modern contrast compression therapy enhances this principle by combining sequential thermal stimulation with active pneumatic compression. This combination aims to improve not only peripheral circulation but also lymphatic drainage and tissue oxygenation.

Contrast compression therapy has gained popularity in recent years, especially in orthopedic and sports rehabilitation, due to its potential benefits in controlling pain and edema. Technological advancements have enabled these systems to deliver precisely regulated temperature, pressure, and treatment durations, allowing for a more controlled and personalized approach compared to conventional methods. Despite promising results in musculoskeletal applications, no clinical trial to date has specifically evaluated the effects of contrast compression therapy in the neurological rehabilitation context, particularly for patients with post-stroke CRPS.

Therefore, this randomized controlled trial was designed to investigate whether adding contrast compression therapy to conventional rehabilitation provides additional benefits for pain control, edema reduction, functional recovery, and motor improvement in patients diagnosed with post-stroke CRPS, aiming to address an important gap in the current literature.

ELIGIBILITY:
Inclusion Criteria:

* Age between 25 and 80 years
* First-ever stroke diagnosed within the previous 12 months
* Diagnosis of upper-extremity complex regional pain syndrome type I (CRPS-I) according to the Budapest clinical criteria
* Subacute-stage CRPS affecting the upper limb
* Mini-Mental State Examination (MMSE) score greater than 23
* Provided written informed consent

Exclusion Criteria:

* Unstable medical condition
* Hemispatial neglect
* Sensory or motor aphasia
* Shoulder subluxation
* CRPS due to causes other than stroke
* Bilateral CRPS-I
* History of psychotic disorder
* Coexisting neuropathic pain syndromes (e.g., diabetic neuropathy)
* Presence of open wounds in the treatment area

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-01-09 (Actual); Study Completion 2023-01-09 (Actual)

PRIMARY OUTCOMES:
Change in Pain Intensity | Baseline and after 4 weeks of treatment
  Upper extremity pain will be assessed at rest and during activity using the Visual Analog Scale.
Change in Upper Extremity Edema Volume | Baseline and after 4 weeks of treatment
  Edema will be measured by the water displacement method using a hand volumeter.

SECONDARY OUTCOMES:
Change in Clinical Motor Recovery | Baseline and after 4 weeks of treatment
  Motor recovery will be evaluated using the Brunnstrom Motor Recovery Stages for the upper extremity and hand.
Change in Neuropathic Pain Probability | Baseline and after 4 weeks of treatment
  Neuropathic pain probability will be assessed using the painDETECT Questionnaire.
Change in Spasticity | Baseline and after 4 weeks of treatment
  Spasticity will be measured using the Modified Ashworth Scale.
Change in Functional Independence | Baseline and after 4 weeks of treatment
  Functional status will be assessed using the motor subscale of the Functional Independence Measure.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD due to patient confidentiality and ethical restrictions.

REFERENCES:
- [Derived] Akinci MG, Polat CS, Tombak Demircakan A, Bukun YZ, Dalyan M. Effectiveness of contrast compression therapy for post-stroke complex regional pain syndrome: a randomized control trial. Top Stroke Rehabil. 2025 Nov 19:1-10. doi: 10.1080/10749357.2025.2589193. Online ahead of print. PMID 41261073